CLINICAL TRIAL: NCT07254312
Title: Correlation of Venetoclax Plasma Concentrations With Toxicity of Hypometilating Agents and Venetoclax Combination for Acute Myeloid Leukemia Patients in Remission.
Acronym: VEN-AML
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Patrizia Zappasodi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: VEN-AML
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-03

CONDITIONS: AML (Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Venetoclax (VEN) is a potent and selective oral inhibitor of the BCL-2 gene and has shown anti-leukemic activity when used in combination with hypomethylating agents (HMA) in patients with Acute Myeloid Leukemia (AML), both newly diagnosed and in relapse or refractory (R/R) stages. A daily dose of 400 mg has shown the best results in terms of efficacy, toxicity, and low early mortality rates (DiNardo et al., Blood 2019). The HMA-VEN combination has been approved for the treatment of newly diagnosed AML patients who are not candidates for intensive therapy. However, although this treatment is considered low-intensity, it causes a non-negligible toxicity profile, especially hematological toxicity, even in patients who have already achieved remission. As a result, treatment often needs to be interrupted, and VEN dosage adjusted in subsequent cycles.

An analysis by Pratz et al. (Pratz et al., Am J Hematol 2022) following the publication of the pivotal trial reported grade IV cytopenias lasting at least 7 days in the cycles following remission in 161 (87%) patients in the VEN+Azacitidine arm. Furthermore, plasma concentrations of VEN were analyzed in patients who developed grade IV cytopenias for at least 7 days, and no correlation was found between VEN plasma levels and the number of observed cytopenias.

In the routine management of these patients, when hematologic toxicity occurs, the approach varies greatly from center to center and is based on the individual experience and assessment of the referring clinician. As a result, there is no standardized approach. Plasma concentrations of VEN are not routinely measured during treatment.

A better understanding of the factors determining the variable toxicity observed in patients in remission could optimize treatment to improve patient tolerability and allow for the regular administration of therapy, which is essential for maintaining leukemia remission status.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed Acute Myeloid Leukemia treated with HMA-VEN in disease remission (from the first post-remission cycle).

Exclusion Criteria:

* undergoing treatment with moderate or strong Cytochrome 3A4 inhibitors or inducers,
* unwilling to receive treatment as previously specified and to be tested for VEN plasma levels at the previously specified timepoint.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study population: patients with newly diagnosed Acute Myeloid Leukemia treated with HMA-VEN in disease remission (from the first post-remission cycle).
  Patients will be excluded if they are undergoing treatment with moderate or strong Cytochrome 3A4 inhibitors or inducers, or if they are unwilling to receive treatment as previously specified and to be tested for VEN plasma levels at the previously specified timepoint.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Analysis of the association between VEN plasma levels and the incidence of grade IV neutropenia. | 18 months
  Venetoclax plasma concentrations are determined by liquid chromatography coupled to mass spectrometry. The method was developed and validated according to the European Medicines Agency (EMA) guidelines. The drug is separated from the matrix by protein precipitation obtained by adding an acidified solution (0.1% HCOOH: 0.1%) of acetonitrile/methanol in a 1:1 ratio (200 µL) to the test samples (50 µL). The deuterated analogue, Venetoclax-D7, was chosen as the internal standard (IS). The analyte and IS are ionized with an ESI (Electrospray Ionization) source in positive mode. The observed mass transitions are m/z 868.1 > 320.7; 635.5 and m/z 875.2 > 320.8; 642.9 for Venetoclax and IS, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Oncologia, Pavia, Pavia, Italy